CLINICAL TRIAL: NCT03290391
Title: Linking Infectious and Narcology Care-Part II
Acronym: LINC-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-36706; R01DA045547 (NIH)
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: HIV Infection; Drug Use
Keywords: Russia; Substance use; Peer case managers; ART; HIV
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Drug Therapy; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LINC-II (Experimental): LINC-II is a multi-faceted intervention combining pharmacological therapy (i.e., ART and naltrexone for opioid use disorder) and 12 months of strengths-based case management delivered to coordinate care across the narcology and HIV health care systems.
  Interventions: Other: Rapid ART initiation; Drug: Pharmacotherapy for opioid use disorder; Behavioral: Strengths-based HIV case management
- Standard of Care (No Intervention): Participants randomized to the control group will receive the narcology hospital's standard of care, which is detoxification with or without stabilization. Prior to discharge, those identified as HIV-infected are given contact details for an HIV clinic, not an appointment. Upon discharge, patients are encouraged to receive outpatient narcology treatment, monthly, for 1 year. For this study, with regard to linkage to HIV medical care, patients will be given printed information about where to obtain HIV medical care and a resource card containing harm reduction information.

INTERVENTIONS:
Other: Rapid ART initiation — The infectionist will streamline the approval with the ultimate goal of starting participants on ART while they are still hospitalized at the City Addiction Hospital.
  Arms: LINC-II
Drug: Pharmacotherapy for opioid use disorder — Thirteen months of naltrexone treatment for opioid use disorder (injection at baseline, followed by 4 implants).
  Other Names: Naltrexone
  Arms: LINC-II
Behavioral: Strengths-based HIV case management — Strengths-based case management: 10 sessions over 12 months in which a trained case manager (CM) meets individually with patients to motivate them to engage in HIV medical care by supporting the recognition of their own strengths to make positive changes in their lives and ultimately improve their HIV outcomes.
  Arms: LINC-II

SUMMARY:
This study, "Linking Infectious and Narcology Care - Part II (LINC-II)," will implement and evaluate a multi-faceted intervention (LINC-II), via a two-armed randomized controlled trial among 240 HIV-infected PWID in St. Petersburg. LINC-II, comprised of pharmacological therapy (i.e., rapid access to ART and receipt of naltrexone for opioid use disorder) and 12 months of strengths-based case management, will assess HIV outcomes (e.g., HIV viral load suppression), impact on care systems and cost-effectiveness of the intervention.

DETAILED DESCRIPTION:
Russia and Eastern Europe continue to have one of the fastest growing HIV epidemics in the world, with highest transmission risks among people who inject drugs (PWID) and their sexual partners. While routine HIV testing within addiction treatment systems in Russia (i.e., narcology hospitals) is the norm, links between the narcology and HIV care systems are limited and ineffective. In St. Petersburg 50-60% of PWID are HIV-infected, yet among this population less than 10% are on antiretroviral therapy (ART). For Russia to make progress toward the UNAIDS 90-90-90 targets (i.e., 90% aware of HIV diagnosis, 90% of those diagnosed on ART and 90% of those on ART with suppressed HIV viral load [HVL]), a bold new strategy is required. The objective of this study, "Linking Infectious and Narcology Care - Part II (LINC-II)," is to implement and evaluate, via a two-armed randomized controlled trial among 240 HIV-infected PWID, a multi-faceted intervention combining pharmacological therapy (i.e., rapid access to ART and receipt of naltrexone for opioid use disorder) and 12 months of strengths-based case management.

The central hypothesis is that LINC-II will lead to marked progress toward the achievement of the 90-90-90 HIV cascade of care targets among HIV-infected PWID, relative to current standard of care, and that LINC-II will facilitate health system coordination of narcology and HIV care. LINC-II aims to: 1) evaluate the effectiveness of LINC-II on undetectable HVL at 12 months (primary outcome), initiation of ART within 28 days of randomization, change in CD4 count from baseline to 12 months, retention in HIV care (i.e., ≥ 1 visit to medical care in 2 consecutive 6 month periods), and undetectable HVL at 6 months; 2) evaluate the impact of LINC-II on coordinated care across the narcology and HIV health care systems, using mixed methods data from health care providers, administrators, and patients; and 3) evaluate the cost-effectiveness of the intervention to inform policy makers on scaling up the LINC-II approach both within Russia and other countries with HIV epidemics driven by injection drug use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* HIV infected
* Hospitalized at narcology hospital
* History of injection drug use
* Current diagnosis of opioid use disorder
* Provision of information for 2 contacts to assist with follow-up
* Address within 100 kilometers of St. Petersburg
* Possession of a telephone (home or cell)
* Able and willing to comply with all study protocols and procedures

Exclusion Criteria:

* Not fluent in Russian
* Cognitive impairment
* Pregnancy, planning to become pregnant, or breastfeeding
* ART use in past 30 days prior to hospitalization
* Known hypersensitivity to naltrexone
* Acute severe psychiatric illness (i.e. ,answered yes to any of the following: past three month active hallucinations; mental health symptoms prompting a visit to the ED or hospital; mental health medication changes due to worsening symptoms; presence of suicidal ideations)
* Known history of liver failure
* ALT or AST >5 times the upper limit of normal
* Known severe thrombocytopenia (<50k)
* Known coagulation disorder/taking anticoagulation medications
* Body habitus that precludes intramuscular injection
* Known hypersensitivity to naloxone
* Known history of Raynaud's disease
* Known history of Itsenko-Cushing syndrome
* Known history of generalized mycoses
* Known history of glaucoma
* Known history of osteoporosis.
* Planned surgeries in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Samet, MD MA MPH, Principal Investigator — Boston University
Locations (2):
- Russia (2):
  - First St. Petersburg Pavlov State Medical University, Saint Petersburg
  - City Addiction Hospital, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosen S, Blokhina E, Truong V, Bereznicka A, Gnatienko N, Quinn E, Lioznov D, Krupitsky E, Michals A, Lunze K, Samet JH. Comparative costs and potential affordability of a multifaceted intervention to improve treatment outcomes among people with HIV who inject drugs in Russia: economic evaluation of the LINC-II randomized controlled trial. J Int AIDS Soc. 2024 Feb;27(2):e26208. doi: 10.1002/jia2.26208. PMID 38403887
- [Derived] Samet JH, Blokhina E, Cheng DM, Rosen S, Lioznov D, Lunze K, Truong V, Gnatienko N, Quinn E, Bushara N, Raj A, Krupitsky E. Rapid access to antiretroviral therapy, receipt of naltrexone, and strengths-based case management versus standard of care for HIV viral load suppression in people with HIV who inject drugs in Russia (LINC-II): an open-label, randomised controlled trial. Lancet HIV. 2023 Sep;10(9):e578-e587. doi: 10.1016/S2352-3018(23)00143-1. PMID 37659841
- [Derived] Bovell-Ammon BJ, Kimmel SD, Cheng DM, Truong V, Michals A, Vetrova M, Hook K, Idrisov B, Blokhina E, Krupitsky E, Samet JH, Lunze K. Incarceration history, antiretroviral therapy, and stigma: A cross-sectional study of people with HIV who inject drugs in St. Petersburg, Russia. Int J Drug Policy. 2023 Jan;111:103907. doi: 10.1016/j.drugpo.2022.103907. Epub 2022 Nov 17. PMID 36402082
- [Derived] Gnatienko N, Lioznov D, Raj A, Blokhina E, Rosen S, Cheng DM, Lunze K, Bendiks S, Truong V, Bushara N, Toussova O, Quinn E, Krupitsky E, Samet JH. Design of a randomized controlled trial to Link Infectious and Narcology Care (LINC-II) in St. Petersburg, Russia. Addict Sci Clin Pract. 2020 Jan 13;15(1):1. doi: 10.1186/s13722-020-0179-8. PMID 31931884

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 953 potential participants were assessed for eligibility via medical record pre-screen. 642 were ineligible and 75 did not proceed with in-person screener due to being previously enrolled or discharged early.
  236 potential eligible participants completed the in-person screener; 7 did not meet the inclusion criteria and 4 declined to participate. 225 completed the baseline interview and were randomized.
Period: Allocation
Arm/Group | LINC-II | Standard of Care
Started | 111 | 114
Completed | 111 | 114
Not Completed | 0 | 0
Period: Completed 6 Month Assessment
Arm/Group | LINC-II | Standard of Care
Started | 111 | 114
Completed | 79 | 85
Not Completed | 32 | 29
Period: Completed 12 Month Assessment
Arm/Group | LINC-II | Standard of Care
Started | 111 | 114
Completed | 82 | 83
Not Completed | 29 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LINC-II | Standard of Care | Total
Number analyzed (Participants) | 111 | 114 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (5) | 37 (5) | 37 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 42 | 89
  Male | 64 | 72 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 111 | 114 | 225
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 110 | 113 | 223
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 111 | 114 | 225

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HIV Viral Load at 12 Months
Description: Number of participants with undetectable HIV viral load at 12 months, assessed by HIV viral load lab test (<40 copies per milliliter)
Time Frame: 12 months post randomization
Population: Participants were analyzed according to the intention-to-treat principle. Missing data was accounted for with multiple imputations (using 25 generated complete datasets).
Measure: Number; unit: percentage of participants
Arm/Group | LINC-II | Standard of Care
Number analyzed (Participants) | 111 | 114
percentage of participants | 46.9 | 22.7

2. Secondary Outcome: Initiation of Antiretroviral Therapy (ART)
Description: Number of participants who initiated ART within 28 days of randomization. Data will be extracted from medical record.
Time Frame: Within 28 days of randomization
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LINC-II | Standard of Care
Number analyzed (Participants) | 111 | 114
percentage of participants | 73.9 | 11.4

3. Secondary Outcome: Change in Mean CD4 Count From Baseline to 12 Months
Description: The change in the mean CD4 count (CD4 cells per cubic millimeter) will be calculated from the baseline and 12 months lab results
Time Frame: Change from baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | LINC-II | Standard of Care
Number analyzed (Participants) | 111 | 114
cells per cubic millimeter | 56 (171) | -8 (193)

4. Secondary Outcome: Retention in HIV Care
Description: Number of participants who had at least 1 visit to HIV medical care in 2 consecutive 6 month periods. Data will be extracted from medical record.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LINC-II | Standard of Care
Number analyzed (Participants) | 111 | 114
percentage of participants | 51.4 | 35.1

5. Secondary Outcome: Undetectable HIV Viral Load at 6 Months
Description: Number of participants with undetectable HIV viral load at 6 months, assessed by HIV viral load lab test (<40 copies per milliliter).
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LINC-II | Standard of Care
Number analyzed (Participants) | 111 | 114
percentage of participants | 35.4 | 12.9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of the 12-month study period.
Arm/Group | LINC-II | Standard of Care
All-Cause Mortality (participants affected / at risk) | 4/111 | 10/114
Serious Adverse Events (participants affected / at risk) | 9/111 | 13/114
Other Adverse Events (participants affected / at risk) | 13/111 | 3/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LINC-II (N=111) | Standard of Care (N=114)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Death due to overdose (Social circumstances) | 3 (3) | 2 (2)
Death due to heart failure (Cardiac disorders) | 1 (1) | 3 (3)
Death due to suicide (Social circumstances) | 0 (0) | 1 (1)
Death due to sepsis (Infections and infestations) | 0 (0) | 1 (1)
Death due to COVID (Infections and infestations) | 0 (0) | 2 (2)
Death due to acute alcohol intoxication (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LINC-II (N=111) | Standard of Care (N=114)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
General weakness (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elevated AST (Investigations) | 4 (4) | 0 (0)
Elevated ALT (Investigations) | 1 (1) | 0 (0)
Wound infection (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT03290391/Prot_SAP_001.pdf
  • Informed Consent Form (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT03290391/ICF_000.pdf